CLINICAL TRIAL: NCT04390009
Title: Exploratory Study of Entire-body PET Scans for Multiple Sclerosis
Brief Title: Entire-body PET Scans for Multiple Sclerosis
Acronym: EPSMS
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Brain Health Alliance (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: BHA-2020-11
Record Dates: First submitted 2020-05-12; First posted 2020-05-15 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Entire-body PET imaging
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Different PET-CT scanners (make and model) determine the different study arms for the intervention defined as a PET-CT medical imaging scan with the Amyvid imaging agent.
Masking Description: Participants will be de-identified; results will be anonymized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Siemens Biograph Vision PET-CT scans (Other): Parallel study arms defined by PET-CT scanners by different manufacturer and model
  Interventions: Diagnostic Test: Entire-body PET-CT scans; Drug: Amyvid radiopharmaceutical
- United Imaging uEXPLORER PET-CT scans (Other): Parallel study arms defined by PET-CT scanners by different manufacturer and model
  Interventions: Diagnostic Test: Entire-body PET-CT scans; Drug: Amyvid radiopharmaceutical

INTERVENTIONS:
Diagnostic Test: Entire-body PET-CT scans — Entire-body PET-CT scans will be performed with state-of-the-art scanners with different manufacturers' models including Siemens Biograph Vision, United Imaging uEXPLORER and possibly other recently FDA-approved PET-CT scanners.
Drug: Amyvid radiopharmaceutical — Amyvid (F18-florbetapir) will be evaluated for binding to white matter of the peripheral and central nervous system of participants

SUMMARY:
To evaluate whether an entire-body positron emission tomography (PET) scanner can be exploited to improve evaluation, monitoring and measurement of both peripheral and central demyelination in multiple sclerosis (MS) patients.

DETAILED DESCRIPTION:
To collect exploratory data using the most recent PET-CT scanners with their increased detection sensitivity and spatial resolution for the evaluation of F18-florbetapir radiopharmaceutical uptake in the nervous system of the entire body with special attention to correlation of radiotracer activity levels in the myelinated, demyelinated, or remyelinated white matter of multiple sclerosis (MS) patients compared to normal healthy subjects. The pilot study will be conducted on 20 participants as a clinical research trial of PET amyloid and myelin imaging with the primary objective of identifying possible differences in F18-florbetapir radiotracer activity for MS patients compared to normal healthy subjects, and the secondary objective of monitoring psychological health of those participants who elect to be informed of imaging results and who complete a panel of psychometric scales before and after imaging results disclosure.

ELIGIBILITY:
Inclusion Criteria:

* Multiple sclerosis (MS) patients diagnosed by a credentialed neurologist experienced with care of multiple sclerosis patients.
* Normal healthy subjects.
* Willing and able to lie motionless on the PET-CT scanner bed for at least 10 minutes and up to 20 minutes for the duration of the PET-CT medical imaging scan.

Exclusion Criteria:

* Any additional complicating medical illness other than MS including any other neuropsychiatric illness unrelated to MS diagnosed prior to the onset of initial symptoms of MS.
* Pregnancy or breast feeding.
* Diabetes or other metabolic-endocrine disorders.
* Any known concomitant acute infection.
* History of metastatic or locally invasive cancer.
* Recent surgery, chemotherapy or radiation therapy.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Entire-body PET imaging of demyelination of peripheral and central nervous system | During 1 day single PET-CT scan
  Exploratory analysis of relative regional increases and/or decreases of Amyvid activity
Psychometric questionnaire for monitoring psychological health | Up to 90 days
  Assessments of participants

CONTACTS AND LOCATIONS:
Overall Officials: Carl Taswell, MD, PhD, Principal Investigator — Brain Health Alliance
Locations (1):
- Brain Health Alliance, Ladera Ranch, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All information and data will be shared with investigators at collaborating imaging sites prior to publication of the results, and with all other investigators after publication of the results.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Anonymized de-identified data will be available after completion of the study.
Access Criteria: Anonymized de-identified data will be available to registered users of the data.
URL: https://epsms.brainhealthalliance.net

REFERENCES:
- [Background] Taswell C, Villemagne VL, Yates P, Shimada H, Leyton CE, Ballard KJ, Piguet O, Burrell JR, Hodges JR, Rowe CC. 18F-FDG PET Improves Diagnosis in Patients with Focal-Onset Dementias. J Nucl Med. 2015 Oct;56(10):1547-53. doi: 10.2967/jnumed.115.161067. Epub 2015 Aug 6. PMID 26251415
- See also: Research Protocol for Exploratory Study of Entire-body PET Scans for Multiple Sclerosis (EPSMS) — https://www.brainiacsjournal.org/arc/pub/Taswell2020EPSMS
- See also: Amended Protocol for Exploratory Study of Entire-body PET Scans for Multiple Sclerosis (EPSMS) — https://www.brainiacsjournal.org/arc/pub/Taswell2023EPSMS
- See also: EPSMS Clinical Trial — https://epsms.brainhealthalliance.net/